CLINICAL TRIAL: NCT05582148
Title: Meniere Disease and Hearing Aids
Acronym: MMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC22.0289
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Meniere Disease; Hearing Loss, Sensorineural
MeSH Terms: conditions — Meniere Disease; Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: cohort followed up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Hearing aids fitting — Fitting hearing aids and evaluating the results at 6 months

SUMMARY:
Patients with unilateral Meniere Disease often a distortion that causes difficulties to provide hearing aids to these patients. Those patients have two main problems: disorders in noise comprehension due to interaural threshold difference and increase in the distortion during dizziness crisis.

Due to these problems, some people cannot be fitting with hearing aids because the compression needed is too high or the discomfort in noise is not bearable for patients.

Our aim is to evaluate and to propose a way to adjust hearing aids to restore binaural hearing with comfort.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 y.o
* Meniere disease as define by the Barany Society
* Unilateral deafness with a threshold over 50dB
* Normal ear with a threshold above 30dB
* Interaural threshold difference of at least 30dB
* Patient who has already an hearing aids and satisfied with it

Exclusion Criteria:

* Absence of consent of the patient or not able to give it
* Patient with hearing aids well fitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the comprehension in noise | 6 months
  Evaluation with the FrMatrix test of the noise comprehension at 6 months

SECONDARY OUTCOMES:
Correlation between the ear recruitment and the settings of the hearing aids | 6 months
  Correlation between the fowler test and the MPO modifications

CONTACTS AND LOCATIONS:
Overall Officials: Ashley BAGUANT, Principal Investigator — University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cubick J, Buchholz JM, Best V, Lavandier M, Dau T. Listening through hearing aids affects spatial perception and speech intelligibility in normal-hearing listeners. J Acoust Soc Am. 2018 Nov;144(5):2896. doi: 10.1121/1.5078582. PMID 30522291
- [Result] Havia M, Kentala E, Pyykko I. Hearing loss and tinnitus in Meniere's disease. Auris Nasus Larynx. 2002 Apr;29(2):115-9. doi: 10.1016/s0385-8146(01)00142-0. PMID 11893444
- [Result] Hood JD. Speech discrimination in bilateral and unilateral hearing loss due to Meniere's disease. Br J Audiol. 1984 Aug;18(3):173-7. doi: 10.3109/03005368409078945. PMID 6487852
- [Result] McNeill C, McMahon CM, Newall P, Kalantzis M. Hearing aids for Meniere's syndrome: implications of hearing fluctuation. J Am Acad Audiol. 2008 May;19(5):430-4. doi: 10.3766/jaaa.19.5.5. PMID 19253813
- [Result] Sato G, Sekine K, Matsuda K, Ueeda H, Horii A, Nishiike S, Kitahara T, Uno A, Imai T, Inohara H, Takeda N. Long-term prognosis of hearing loss in patients with unilateral Meniere's disease. Acta Otolaryngol. 2014 Oct;134(10):1005-10. doi: 10.3109/00016489.2014.923114. Epub 2014 Jul 16. PMID 25029391
- [Result] Valente M, Mispagel K, Valente LM, Hullar T. Problems and solutions for fitting amplification to patients with Meniere's disease. J Am Acad Audiol. 2006 Jan;17(1):6-15. doi: 10.3766/jaaa.17.1.2. PMID 16640056